CLINICAL TRIAL: NCT06320522
Title: Characterizing the Influence of Exogenous Ketosis on Circulating and Hepatic Metabolism in a Postprandial and Postabsorptive State in Adults Free From Metabolic Disease
Brief Title: Exogenous Ketosis in a Fed and a Fasted State
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: R82053/RE002
Record Dates: First submitted 2024-03-05; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Ketosis; Exogenous Ketosis
Keywords: Exogenous Ketosis; Hepatic; Metabolism; Postprandial; Postabsorptive
MeSH Terms: conditions — Ketosis | interventions — rVSV-deltaG-spike COVID-19 vaccine; (R)-3-hydroxybutyl (R)-3-hydroxybutyrate; sucrose octaacetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fed - Ketone Monoester (Active Comparator): Ketone monoester drink (573 mg∙kg-1 body weight) provided 1 hour after a 2 g∙kg-1 bodyweight of carbohydrate mixed nutrient breakfast meal
  Interventions: Dietary Supplement: Ketone Monoester
- Fed - Placebo (Placebo Comparator): Placebo drink provided 1 hour after a 2 g∙kg-1 bodyweight of carbohydrate mixed nutrient breakfast meal
  Interventions: Dietary Supplement: Placebo
- Fasted - Ketone Monoester (Active Comparator): Ketone monoester drink (573 mg∙kg-1 body weight) provided whilst fasted
  Interventions: Dietary Supplement: Ketone Monoester
- Fasted - Placebo (Placebo Comparator): Placebo drink provided whilst fasted
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone Monoester — Commercial dietary supplement intended raise blood ketone body levels
  Other Names: deltaG; (R)-3-hydroxybutyl (R)-3-hydroxybutyrate
  Arms: Fasted - Ketone Monoester; Fed - Ketone Monoester
Dietary Supplement: Placebo — Placebo drink (2mM sucrose octaacetate) taste and volume matched to the ketone monoester drinks
  Other Names: Sucrose Octaacetate
  Arms: Fasted - Placebo; Fed - Placebo

SUMMARY:
The kinetics of circulating βHB following ingestion of the ketone monoester are dependent on several variables that determine the balance between appearance into, and disappearance from, the bloodstream. These dynamics have been well characterised in fasted humans but in the real world the ketone monoester is likely to be ingested in a fed state, pertinently within athletic spheres consumption would proceed a substantial high-carbohydrate meal. Within this, it is unclear how metabolism under exogenous ketosis might be affected in a fed versus fasted state.

This four-arm crossover study looks to characterise the relationship between feeding status, βHB pharmacokinetics, and resting metabolism.

As exogenous ketosis is known to reduce circulating glucose levels, this study will also explored if hepatic metabolism - for example, de novo lipogenesis - might consequently be altered, with implications for metabolic disease states such as Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) and type II diabetes.

Participants will be asked to consume either the ketone monoester drink or a placebo drink when fasted and when having previously consumed a meal.

DETAILED DESCRIPTION:
Adults free from metabolic disease will be recruited for this randomised-counterbalanced crossover study. Participants will attend four study visits.

Participants will consume a prescribed isocaloric high-carbohydrate diet for two days prior to each visit to standardise dietary intake.

For two of these visits participants will remain 'fasted' throughout, and for the two 'fed' visits they will consume a mixed-nutrient breakfast meal. The breakfast for the 'fed' visits will provide 2g∙kg-1 bodyweight of carbohydrate.

Heavy water (D2O) will be consumed the evening preceding, and during, each fed study visit to achieve ~0.4% plasma enrichment, in order to quantify the contribution of hepatic de novo lipogenesis to VLDL-TG.

At these visits they will consume either a ketone monoester (KME) or taste/volume-matched placebo (PLA) drink. The nature of this drink will be single blinded and consumed after the breakfast meal during the 'fed' visits.

Therefore the four visits will be as follows: fed-KME, fed-PLA, fasted-KME, fasted-PLA.

Blood and breath samples will be collected at fasting and across a 6 hour period after consuming the KME or PLA drink. Subjective measures of gastrointestinal distress and appetite will also be assessed.

This study aims to establish how feeding state might affect the appearance of βHB into the bloodstream, circulating metabolism, and hepatic metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Habitually consuming a mixed macronutrient diet
* Fluent in English, no communication impairments, willing & able to give informed consent for participation in the study
* Not currently taking any medication (except the contraceptive pill)
* No food allergies incompatible with the supplement drinks or with the standardised breakfast where a suitable substitution cannot be practically made
* Female-only - on contraception (pill/implant/coil/etc); not pregnant/currently breastfeeding; pre-menopausal; not undertaking hormone replacement therapy (HRT)
* In the investigator's opinion - able and willing to comply with all study requirements

Exclusion Criteria:

* Significant cardiovascular disease or metabolic risk factors, or family history of it, on health screening questionnaire
* Food allergies incompatible with the supplement drinks or standardised breakfast
* Having been on a ketogenic diet in the 6 months prior to enrolment
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study/the participant's ability to participate in the study
* Concurrently a participant in any other dietary intervention study/have taken part in one within 1 month of enrolment
* Diabetic
* Pregnant or breastfeeding
* Known history of moderate-to-severe motion sickness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Plasma β-hydroxybutyrate (βHB) kinetics | 7 hours (fasted arrival through to 6 hours after consumption of the KME or PLA drink)
  Changes in concentration of plasma βHB (mM) over the post-drink time period
Plasma glucose kinetics | 7 hours (fasted arrival through to 6 hours after consumption of the KME or PLA drink)
  Changes in concentration of plasma glucose (mM) over the post-drink time period
Postprandial de novo lipogenesis (DNL) | 7 hours (fasted arrival through to 6 hours after consumption of the KME or PLA drink)
  DNL in the fed visits - quantified as the incorporation of deuterium from heavy water into newly synthesised palmitate within very low-density lipoprotein-triglyceride (VLDL-TG)

SECONDARY OUTCOMES:
Plasma biochemistry | 7 hours (fasted arrival through to 6 hours after consumption of the KME or PLA drink)
  Changes in concentration of plasma lactate, insulin, nonesterified fatty acid (NEFA), triglyceride (TG), glycerol, and urea (all mM) over the post-drink time period
Very low-density lipoprotein-triglyceride (VLDL-TG) fatty acid composition | 7 hours (fasted arrival through to 6 hours after consumption of the KME or PLA drink)
  Changes in fatty acid composition (mol%) of VLDL-TG over the post-drink time period
Breath acetone | 7 hours (fasted arrival through to 6 hours after consumption of the KME or PLA drink)
  Changes in concentration of breath acetone (arbitrary units) over the post-drink time period
Urine volume | 7 hours (fasted arrival through to 6 hours after consumption of the KME or PLA drink)
  Volume (ml) of urine over the post-drink time period
Urine composition | 7 hours (fasted arrival through to 6 hours after consumption of the KME or PLA drink)
  βHB concentration (mM) of urine over the post-drink time period
Indirect calorimetry | 7 hours (fasted arrival through to 6 hours after consumption of the KME or PLA drink)
  Changes in Respiratory Quotient (RQ; unitless) over the post-drink time period
Subjective measures of appetite | 7 hours (fasted arrival through to 6 hours after consumption of the KME or PLA drink)
  Changes in perceptions of appetite over the post-drink period Appetite sensations will be assessed using a validated 10-point visual analogue scale (score: 0 - minimal, 10 - maximal) which will be presented to participants on printed paper This posed four questions - "How hungry do you feel?", "How full do you feel?", "How satisfied do you feel?", and "How much do you think you can eat now?"
Subjective measures of gastrointestinal distress | 7 hours (fasted arrival through to 6 hours after consumption of the KME or PLA drink)
  Changes in perceptions of gastrointestinal (GI) distress over the post-drink period GI distress will be assessed using a literature-standard 0-8 Likert scale questionnaire quantified at upper abdominal (reflux, bloating, nausea, vomiting), lower abdominal (cramps, flatulence, abdominal pain, diarrhoea), and systemic (dizziness, headache, muscle cramp, urge to urinate) levels (severity score: 0 - minimal, 8 - maximal)

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Centre for Diabetes, Endocrinology, and Metabolism (OCDEM), Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No